CLINICAL TRIAL: NCT06562530
Title: High Tone Power Therapy Versus Transcutaneous Electrical Nerve Stimulation on Spasticity and Selected Kinematic Gait Parameters in Stroke Patients
Brief Title: Effect of High Tone Power Therapy on Spasticity and Gait Kinematics in Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jasmine Magdy Mahmoud Abd-elkhalik, lecturer assistant of physical therapy for neurology and neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P. T. REC/012/004855
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: high tone power therapy; spatiotemporal gait parameters; gait kinematics
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT). True experimental research design study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (Active Comparator): 15 patients: receiving 36 sessions of selected physical therapy program for 1 hour 3 times per week for 3 months.
  Interventions: Other: selected physical therapy program
- The study group1 (Experimental): 15 patients: receiving 36 sessions of High tone power therapy program for 30 minutes and selected physical therapy program for 30 minutes 3 times per week for 3 months (total session: 1 hour).
  Interventions: Device: high tone power therapy; Other: selected physical therapy program
- The study group 2 (Experimental): 15 patients: receiving 36 sessions of TENS program for 30 minutes and selected physical therapy program for 30 minutes 3 times per week for 3 months (total session: 1 hour).
  Interventions: Device: transcutaneous electrical nerve stimulation (TENS); Other: selected physical therapy program

INTERVENTIONS:
Device: high tone power therapy — sessions are applied for 30 minutes, 3 times per week, for 3 months
  Arms: The study group1
Device: transcutaneous electrical nerve stimulation (TENS) — sessions are applied for 30 minutes, 3 times per week, for 3 months
  Arms: The study group 2
Other: selected physical therapy program — sessions are applied for 1 hour, 3 times per week, for 3 months in form o fstretching exercise , range of motion exercises , conventional gait training progressive resistance exercises

SUMMARY:
This study aims to compare between High tone power therapy (modulated frequency current) and Transcutaneous electrical nerve stimulation (fixed frequency current) on spasticity and selected kinematic gait parameters in stroke patients.

DETAILED DESCRIPTION:
Stroke is a neurological deficit attributed to an acute focal injury of the central nervous system (CNS) by a vascular cause . Stroke is one of the leading causes of disability and mortality in the globe, stroke occurs when blood flow to the brain is restricted due to a blocked or ruptured artery; the cerebral energy supply is interrupted, resulting in tissue destruction and widespread neuronal, cognitive impairments, and psychological morbidity .

Stroke is the second major cause of death and disability worldwide with over 13 million new cases annually . Stroke has been described as a major source of both mortality and global disability . Approximately 795,000 people experience stroke annually, and 60% (or 465,000) of them need rehabilitation .

Spasticity is a symptom of stroke, brain and spinal cord damage, multiple sclerosis, cerebral palsy, and other neurological illnesses that cause paralysis . The most common spastic pattern in the lower limbs is adduction and extension of the knee with an Equinovarus foot . This impacts gait patterns and daily functioning activities .

Treatment modalities for the management of spasticity include Stretching, splinting, Neuromuscular electrical stimulation (NMES), extracorporeal shock wave therapy, transcranial and spinal cord magnetic stimulation, Surgical treatment, neurectomy, rhizotomy, and myelotomy; also, many drugs used for treating spasticity oral drugs like Baclofen, Tizanidine, and injectable medications like Phenol/alcohol and Botulinum 2 toxin .

Transcutaneous electrical nerve stimulation (TENS) stimulates large diameter mechano-sensitive nerve fibers in the skin it's a non-invasive treatment that has been reported to affect pain control and sensory stimulation which is commonly used in the treatment of chronic and acute pain with possible mechanisms of action including segmental inhibition, the release of endogenous opioids, counter-irritation, nerve conduction block, increase muscle power and movement function .

High-tone power therapy (HTT) is a unique characteristic of electrotherapy. It uses intermediate frequency, metal-compatible alternating current whose frequency oscillates between approximately 4000 Hz and 33000 Hz, and intensity is adjusted, unlike traditional electrotherapies as transcutaneous electrical nerve stimulation (TENS). Its main effects are introducing energy into the body to activate cells, producing an oscillation or vibration in the cells and tissues to promote metabolism, scattering the mediators of pain and inflammation leading to pain relief, and normalizing cell metabolism and nerve regeneration ).

The effective management of spasticity continues to pose challenges to physiotherapy management, there appears to be a dearth of adequate information on high tone power therapy in the management of spasticity; There are several physiotherapy approaches for managing spasticity but there is a lack of evidence to show which is most effective .

Statement of the problem:

This study will answer the following question: Is there any difference between the effect of high-tone power therapy (modulated frequency current) versus transcutaneous electrical nerve stimulation (fixed frequency current) on spasticity and selected kinematic gait parameters in stroke patients?

ELIGIBILITY:
Inclusion Criteria:

1. Duration of illness not less than six months post-stroke (Hillis A. et al., 2006).
2. Patients' age ranges from forty-five to sixty-five years (Feigin et al., 2022).
3. Body mass index from (18.5 to 24.9).
4. Patients can respond to verbal instructions (Consciousness and orientation to time, place, and person) more than 13 degrees on the Glasco coma scale (Hegazy et al., 2020).
5. Able to walk independently on an even surface without any assistive device (Fan and Yin, 2013).
6. Patients with moderate Spasticity of the ankle joint (grade 2 and 3 According to Modified Ashworth Scale) (Hegazy et al., 2020).

Exclusion Criteria:

1. Subjects with any other Co-existing Progressive neurological disorder (Hegazy et al., 2020).
2. Unstable Cardiac condition (E.g., Acute Myocardial infarction, severe Cardiac Failure) (Teslim et al., 2013).
3. Subjects with any anti-spastic Drugs (Chang et al., 2013).
4. Musculoskeletal disorders affecting gait kinematics such as severe arthritis, knee surgery, and total hip joint replacement, lower limb fractures less than 6 months or contractures of fixed deformity, leg length discrepancy.
5. Any previous Contracture or deformities (Hegazy et al., 2020).
6. Un co-operative patients (Gupta and Chatterjee, 2019).
7. Open wounds, burns, or Loss of sensation (Grevstad et al., 2016).
8. Patients with metal implants (von Lewinski et al., 2009).
9. Visual, auditory problems.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  This scale is used to measure spasticity of Calf muscle in grades from 0 to 5.
Computerized electromyography (EMG) using H/M ratio | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  EMG is an objective device used to measure spasticity of the Soleus muscle in percentage (%)
Ten-meter Walk test(10-MWT) | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  This scale is used to measure walking speed in m/s
  * self-selected walking speed (SSWS) in (m/s).
  * fastest walking speed (FWS) in (m/s).
Time up and go test (TUG) | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  This test is used to measure time taken by patient to apply sit to stand, walk a distance of 3 meters, turn and walk back to the chair in (sec.)
Gait velocity | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  Gait Analyzer Smart Phone Application is an objective tool that assesses gait velocity (m/s).
cadence | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  Gait Analyzer Smart Phone Application is an objective tool that assesses cadence: the number of steps per second in (steps/ s).
step time | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  Gait Analyzer Smart Phone Application is an objective tool that assesses step time in ( msec.)
step time symmetry | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  Gait Analyzer Smart Phone Application is an objective tool that assesses step time symmetry: the symmetry in time between affected and unaffected lower limbs in percentage (%)
step length | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  Gait Analyzer Smart Phone Application is an objective tool that assesses step length by the inertial sensor system symmetry in meters (m).
step length symmetry | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  Gait Analyzer Smart Phone Application is an objective tool that assesses step length symmetry: the symmetry in step length between affected and unaffected lower limbs in percentage (%)

SECONDARY OUTCOMES:
Lafayette Hand-held Dynamometer | measurements will be done 3 days before the start of the treatment program and will be done after 3 days post intervention
  This is an objective device used to measure the isometric contraction of dorsi flexors in pounds (lbs.)

CONTACTS AND LOCATIONS:
Overall Officials: Eman S Fayiz, Professor, Study Chair — Cairo University; Mahmoud Y El-Zanaty, Study Chair — Cairo University; Sandraa M Ahmed, Professor, Study Chair — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No